CLINICAL TRIAL: NCT07068217
Title: Effect of Metronome-Based Structured Rhythmic Exercise Program on Freezing and Gait Parameters in Parkinson Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, merve özel, physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-221
Record Dates: First submitted 2025-07-06; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Parkinson disease; cueing; freezing of gait
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REG (Experimental): Rhythmic Exercise Group: The structured exercise program will be conducted with metronome cues tailored to each participant's cadence using the "Google Metronome" app.
  Both groups will receive a supervised home-based exercise program, overseen via telerehabilitation. Exercises will be performed 3 times per week for 45-60 minutes each session, over 4 weeks (12 sessions total). Progression to the next week's program will require an 80% success rate; otherwise, the same week's program will be repeated. Online supervision will monitor weekly performance.
  Interventions: Other: Exercise
- EG (Active Comparator): Exercise Group: Participants will perform the same exercises at their own pace, without rhythmic cues.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Sample size was determined via G*Power analysis: two groups (n=13 each), total n=26. Participants will be randomized using Random.org into the Rhythmic Exercise Group (REG) or the Exercise Group (EG).
  Both groups will receive a supervised home-based exercise program, overseen via telerehabilitation. Exercises will be performed 3 times per week for 45-60 minutes each session, over 4 weeks (12 sessions total). Progression to the next week's program will require an 80% success rate; otherwise, the same week's program will be repeated. Online supervision will monitor weekly performance.
  Other Names: metronome exercises

SUMMARY:
Background: Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by the loss of dopaminergic neurons in the substantia nigra pars compacta, leading to motor symptoms such as resting tremor, freezing episodes, gait disturbances, rigidity, and bradykinesia. It is estimated that approximately 6.1 million people worldwide live with PD. With disease progression, freezing episodes and gait impairments intensify, significantly limiting independence and increasing both fall risk and mortality. Although a definitive cure is lacking, symptom management relies on pharmacological and non-pharmacological interventions.

In PD patients, adaptability to environmental changes and the ability to process sensory inputs and generate motor responses become impaired. Therefore, sensory re-education using auditory, somatosensory, or visual cues is employed. External cues support motor learning by facilitating initiation and maintenance of movement. By promoting cortical reorganization, these cues can improve gait quality, reduce freezing severity, and enhance participation in daily life.

A commonly used method in this context is Rhythmic Auditory Stimulation (RAS). Administered with metronome beats or music, RAS provides external cues via the auditory system to reorganize gait patterns. In patients experiencing freezing, motor blocks during gait can be overcome through rhythmic stimulation. Numerous studies have reported that RAS improves gait speed, step length, and cadence.

Despite its benefits, there is a paucity of methodologically robust, standardized trials evaluating the effects of RAS on real-world symptoms such as gait disturbances and freezing. Therefore, there is a clear need for structured interventions based on metronome-driven rhythmic cues and clinical trials assessing their impact. Furthermore, investigating feasibility in home settings via telerehabilitation is valuable for enhancing accessibility of such interventions.

Purpose: To assess the effects of a structured rhythmic exercise program using metronome cues on freezing episodes, gait parameters, balance, fall risk, and quality of life in PD patients.

Methods: This randomized controlled trial is planned at Taksim Training and Research Hospital from May 2025 to May 2026. Ethical approval has been granted by Istanbul Medipol University's Non-Interventional Clinical Research Ethics Committee (No. E-10840098-202.3.02-221). Sample size was determined via G*Power analysis: two groups (n=13 each), total n=26. Participants will be randomized using Random.org into the Rhythmic Exercise Group (REG) or the Exercise Group (EG).

Both groups will receive a supervised home-based exercise program, overseen via telerehabilitation. Exercises will be performed 3 times per week for 45-60 minutes each session, over 4 weeks (12 sessions total). Progression to the next week's program will require an 80% success rate; otherwise, the same week's program will be repeated. Online supervision will monitor weekly performance.

REG: The structured exercise program will be conducted with metronome cues tailored to each participant's cadence using the "Google Metronome" app.

EG: Participants will perform the same exercises at their own pace, without rhythmic cues.

At the first visit, the demographic information form containing the demographic information and clinical features of all volunteers will be recorded with the necessary information. Then; The participants' disease severity and disability levels will be assessed with the Unified Parkinson's Disease Rating Scale (UPDRS); Walking parameters such as walking speed, step length, step count, cadence and freezing times during walking will be assessed with the 10-Meter Walk Test (10MYT) using Movemate Version 1; Balance skills will be assessed with the MiniBESTest; Performance, with the Timed Up and Go Test (TUG); Freezing and falls in ADL will be assessed with the Freezing While Walking Scale (WGS) and; Falls, with the International Falls Efficacy Scale (IFES); Quality of life will be assessed with the Parkinson's Disease Quality of Life Questionnaire (PHA-39). The assessment tests will be administered face-to-face at the beginning of the study and at the end of the 4th week, 12-18 hours after taking the medication.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn and Yahr Scale Stage III-IV
* Mini Mental Test Score > 24
* Stable medication use for the last month
* Age range 55-75
* Able to walk 20 meters independently on level ground
* Answering Yes to the first question of the New Freezing of Gait Questionnaire
* Having a caregiver with you during the exercises

Exclusion Criteria:

* Neurological and Orthopedic Disorders Other Than PD
* Medically diagnosed hearing loss
* Patients requiring assistive devices for ambulation
* Dementia
* No internet access via smartphone or computer
* Patients with deep brain pacemakers
* Having vascular lower extremity pathologies
* Not receiving any additional physical therapy during the study period

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
10m Walking Test | week 1 (beginning of study) - week 4 (end of the study)
  10-Meter Walk Test (10MWT) One of the tests recommended by the American Physical Therapy Association Neurology Section as an outcome measure in individuals with PD, the 10MWT is a widely used test to assess walking speed in individuals with walking limitations. In the test, participants are asked to walk at a speed of their own choosing for the normal walking test and as quickly and safely as possible for the fast walking test. Three trials of each test are completed with short rest breaks between trials if necessary. The time for each test is recorded, the average value is calculated and converted to m/s. There are studies in the literature showing that the 10MYT is reliable and valid in individuals with PD.
  In our study, 10MYT will be applied with 'Movemate version 1' and the collected data will be analyzed.
Spatial parameters of walking with Movemate Version 1.0 | week 1 (beginning of the study) - week 2 (end of the study)
  MoveMate Version 1 In this study, the MoveMate Version 1 (*Interrupt Biomedical and Engineering and Joint Stock Company) device will be used to evaluate the spatial parameters of gait in Parkinson's patients. MoveMate Version 1 is a wearable motion tracking system developed for gait analysis, including an accelerometer and gyroscope sensors with a Bosch - BMI270 model IMU (Inertial Measurement Unit) attached to the ankle.
  The device can analyze the patient's gait patterns by recording the patient's gait in real time and store the data securely via a mobile application via Bluetooth connection.
  As part of the study, a 10-m walking test will be applied to the participants by a physiotherapist, and during this process, accelerometer and gyroscope data will be collected in 3 axes with the MoveMate device. The raw data obtained will be analyzed using specially developed software, and basic gait parameters such as step count, step frequency, step length and walking speed will be calculated
Timed Up and Go Test (TUG) | week 1 (beginning of the study)- week 4 (end of the study)
  A simple, widely used and rapid test for assessing mobility, balance and fall risk. To perform the test, participants must get up from a standard chair, walk comfortably to a location 3 meters away from the ground, turn around and return to the chair, and sit back in the same chair. In our study, all steps of the test will be measured in seconds with a stopwatch. The test will be repeated 3 times and the average of these measurements will be analyzed.
MiniBESTest | week 1 (beginning of the study)- week 4 (end of the study)
  It is one of the clinical tests used in the evaluation of walking and balance. It consists of 4 sub-parameters, namely preparatory movement, reactive postural control, sensory orientation, dynamic walking, and a total of 14 items. It is a test that is evaluated over a total of 28 points, requiring an average of 10-15 minutes. High scores indicate high function.
The Freezing of Walking Scale (FWS) | week 1 (beginning of the study- week 4 (end of the study)
  The Freezing of Walking Scale (FWS) was used to determine and evaluate the subjective perception of Parkinson's patients regarding the severity and effect of the degree of freezing on walking performance. This questionnaire consists of 6 questions, 4 of which evaluate the severity of freezing and 2 of which evaluate walking difficulties in general. It is a 5-point scale from 0 to 4, with a total score between 0 and 24. A higher score means that the person's walking performance is more affected by freezing. The validity and reliability study of the FWS in Turkish has been conducted

SECONDARY OUTCOMES:
The International Falls Efficacy Scale (IAES) | week 1 (beginning of the study)- week 4 (end of the study)
  The International Falls Efficacy Scale (IAES) was developed by modifying the Falls Index Scale, which consists of 10 items developed by Tinetti et al. It has been shown to have high test-retest reliability. It evaluates fear of falling during ADL (house cleaning, going up and down stairs, walking, etc.), possible falls, and functional capacity, and consists of 16 items with four answer options. The total score varies between 16 and 64, with a high score indicating a high fear of falling. It has been shown to be reliable and valid in individuals with PD, its internal consistency and test-retest reliability are high, and Visual Analog Scale-Fear of Falling, its validity is moderate-high. The reliability and validity of the Turkish version has been shown in elderly individuals
Parkinson's Disease Quality of Life Questionnaire (PHA-39) | week 1 (beginning of the study)- week 4 (end of the study)
  Parkinson's Disease Quality of Life Questionnaire (PHA-39) It will be used in the assessment of quality of life. PHA-39 is a self-report questionnaire that uses a 5-point Likert scale to assess quality of life such as severity of symptoms of mobility, activities of daily living, emotional well-being, social support, cognition, and communication. The total score ranges from 0 to 100, with higher scores indicating lower quality of life. The validity and reliability study of the questionnaire in Turkish has been conducted.
Unified Parkinson's Disease Rating Scale | week 1-week 4
  UPDRS is considered the gold standard among clinical scales used in the evaluation of Parkinson's disease because it provides comprehensive information in many aspects. UPDRS consists of 4 sections and this scale evaluates; I-Mental state, behavior and mental state (4 questions), II-Daily living activities (13 questions), III-Motor performance (14 questions), IV-Complications of treatment (motor fluctuations, dyskinesias, autonomic dysfunction). The validity and reliability study of the scale has been conducted in Turkish.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medipol Üniversitesi, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ulus Y, Durmus D, Akyol Y, Terzi Y, Bilgici A, Kuru O. Reliability and validity of the Turkish version of the Falls Efficacy Scale International (FES-I) in community-dwelling older persons. Arch Gerontol Geriatr. 2012 May-Jun;54(3):429-33. doi: 10.1016/j.archger.2011.06.010. Epub 2011 Aug 9. PMID 21831462
- [Result] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188
- [Result] Acaröz Candan, S., Çatıker, A., & Özcan, TŞ. Psychometric Properties Of The Turkish Version Of The Freezing Of Gait Questionnaire For Patients With Parkinson's Disease. Neurol Sci Neurophysiol, 2019; 36(1), 44-50.
- [Result] Potter K, Brandfass K. The Mini-Balance Evaluation Systems Test (Mini-BESTest). J Physiother. 2015 Oct;61(4):225. doi: 10.1016/j.jphys.2015.04.002. Epub 2015 Jun 1. No abstract available. PMID 26044345
- [Result] Leddy AL, Crowner BE, Earhart GM. Utility of the Mini-BESTest, BESTest, and BESTest sections for balance assessments in individuals with Parkinson disease. J Neurol Phys Ther. 2011 Jun;35(2):90-7. doi: 10.1097/NPT.0b013e31821a620c. PMID 21934364
- [Result] Huang SL, Hsieh CL, Wu RM, Tai CH, Lin CH, Lu WS. Minimal detectable change of the timed "up & go" test and the dynamic gait index in people with Parkinson disease. Phys Ther. 2011 Jan;91(1):114-21. doi: 10.2522/ptj.20090126. Epub 2010 Oct 14. PMID 20947672
- [Result] Duncan RP, Earhart GM. Remote Delivery of Allied Health Therapies in Parkinson's Disease. J Parkinsons Dis. 2024;14(s1):S219-S226. doi: 10.3233/JPD-230214. PMID 38007673
- [Result] Murgia M, Pili R, Corona F, Sors F, Agostini TA, Bernardis P, Casula C, Cossu G, Guicciardi M, Pau M. The Use of Footstep Sounds as Rhythmic Auditory Stimulation for Gait Rehabilitation in Parkinson's Disease: A Randomized Controlled Trial. Front Neurol. 2018 May 24;9:348. doi: 10.3389/fneur.2018.00348. eCollection 2018. PMID 29910764
- [Result] Avanzino L, Pelosin E, Vicario CM, Lagravinese G, Abbruzzese G, Martino D. Time Processing and Motor Control in Movement Disorders. Front Hum Neurosci. 2016 Dec 12;10:631. doi: 10.3389/fnhum.2016.00631. eCollection 2016. PMID 28018198
- [Result] Ginis P, Nackaerts E, Nieuwboer A, Heremans E. Cueing for people with Parkinson's disease with freezing of gait: A narrative review of the state-of-the-art and novel perspectives. Ann Phys Rehabil Med. 2018 Nov;61(6):407-413. doi: 10.1016/j.rehab.2017.08.002. Epub 2017 Sep 7. PMID 28890341
- [Result] Maidan I, Mirelman A, Hausdorff JM, Stern Y, Habeck CG. Distinct cortical thickness patterns link disparate cerebral cortex regions to select mobility domains. Sci Rep. 2021 Mar 23;11(1):6600. doi: 10.1038/s41598-021-85058-z. PMID 33758214
- [Result] Fasano A, Herman T, Tessitore A, Strafella AP, Bohnen NI. Neuroimaging of Freezing of Gait. J Parkinsons Dis. 2015;5(2):241-54. doi: 10.3233/JPD-150536. PMID 25757831
- [Result] Spildooren J, Vercruysse S, Heremans E, Galna B, Verheyden G, Vervoort G, Nieuwboer A. Influence of Cueing and an Attentional Strategy on Freezing of Gait in Parkinson Disease During Turning. J Neurol Phys Ther. 2017 Apr;41(2):129-135. doi: 10.1097/NPT.0000000000000178. PMID 28263251
- [Result] Martin T, Weatherall M, Anderson TJ, MacAskill MR. A Randomized Controlled Feasibility Trial of a Specific Cueing Program for Falls Management in Persons With Parkinson Disease and Freezing of Gait. J Neurol Phys Ther. 2015 Jul;39(3):179-84. doi: 10.1097/NPT.0000000000000093. PMID 26050074
- [Result] Zhao Y, Nonnekes J, Storcken EJ, Janssen S, van Wegen EE, Bloem BR, Dorresteijn LD, van Vugt JP, Heida T, van Wezel RJ. Feasibility of external rhythmic cueing with the Google Glass for improving gait in people with Parkinson's disease. J Neurol. 2016 Jun;263(6):1156-65. doi: 10.1007/s00415-016-8115-2. Epub 2016 Apr 25. PMID 27113598
- [Result] Suputtitada A, Chen CPC, Pongmala C, Sriyudthsak M, Wilhelm A, Somboon P, Janssen J, Richards J. The Efficacy of a Newly Developed Cueing Device for Gait Mobility in Parkinson's Disease. Parkinsons Dis. 2022 May 18;2022:7360414. doi: 10.1155/2022/7360414. eCollection 2022. PMID 35634541
- [Result] McDonnell P, Rodger M, Teixeira LA, Mitchell G, Doumas M. Sensory reweighting for balance in people living with Parkinson's Disease: Postural adaptation, muscle co-contraction, and perceptual delays. Gait Posture. 2025 Mar;117:342-348. doi: 10.1016/j.gaitpost.2025.01.012. Epub 2025 Jan 14. PMID 39847875
- [Result] Hvingelby VS, Glud AN, Sorensen JCH, Tai Y, Andersen ASM, Johnsen E, Moro E, Pavese N. Interventions to improve gait in Parkinson's disease: a systematic review of randomized controlled trials and network meta-analysis. J Neurol. 2022 Aug;269(8):4068-4079. doi: 10.1007/s00415-022-11091-1. Epub 2022 Apr 5. PMID 35378605
- [Result] Tang L, Zhang L, Liu Y, Li Y, Yang L, Zou M, Yang H, Zhu L, Du R, Shen Y, Li H, Yang Y, Li Z. Optimal dose and type of exercise to improve depressive symptoms in older adults: a systematic review and network meta-analysis. BMC Geriatr. 2024 Jun 7;24(1):505. doi: 10.1186/s12877-024-05118-7. PMID 38849780
- [Result] Yang Y, Wang G, Zhang S, Wang H, Zhou W, Ren F, Liang H, Wu D, Ji X, Hashimoto M, Wei J. Efficacy and evaluation of therapeutic exercises on adults with Parkinson's disease: a systematic review and network meta-analysis. BMC Geriatr. 2022 Oct 21;22(1):813. doi: 10.1186/s12877-022-03510-9. PMID 36271367
- [Result] Song R, Grabowska W, Park M, Osypiuk K, Vergara-Diaz GP, Bonato P, Hausdorff JM, Fox M, Sudarsky LR, Macklin E, Wayne PM. The impact of Tai Chi and Qigong mind-body exercises on motor and non-motor function and quality of life in Parkinson's disease: A systematic review and meta-analysis. Parkinsonism Relat Disord. 2017 Aug;41:3-13. doi: 10.1016/j.parkreldis.2017.05.019. Epub 2017 May 25. PMID 28602515
- [Result] Bryant MS, Rintala DH, Hou JG, Collins RL, Protas EJ. Gait variability in Parkinson's disease: levodopa and walking direction. Acta Neurol Scand. 2016 Jul;134(1):83-6. doi: 10.1111/ane.12505. Epub 2015 Sep 23. PMID 26399376
- [Result] Osborne JA, Botkin R, Colon-Semenza C, DeAngelis TR, Gallardo OG, Kosakowski H, Martello J, Pradhan S, Rafferty M, Readinger JL, Whitt AL, Ellis TD. Physical Therapist Management of Parkinson Disease: A Clinical Practice Guideline From the American Physical Therapy Association. Phys Ther. 2022 Apr 1;102(4):pzab302. doi: 10.1093/ptj/pzab302. PMID 34963139
- [Result] Radder DLM, Ligia Silva de Lima A, Domingos J, Keus SHJ, van Nimwegen M, Bloem BR, de Vries NM. Physiotherapy in Parkinson's Disease: A Meta-Analysis of Present Treatment Modalities. Neurorehabil Neural Repair. 2020 Oct;34(10):871-880. doi: 10.1177/1545968320952799. Epub 2020 Sep 11. PMID 32917125
- [Result] Yoon SY. Update on Parkinson's Disease Rehabilitation. Brain Neurorehabil. 2022 Jul 26;15(2):e15. doi: 10.12786/bn.2022.15.e15. eCollection 2022 Jul. PMID 36743207
- [Result] Simon DK, Tanner CM, Brundin P. Parkinson Disease Epidemiology, Pathology, Genetics, and Pathophysiology. Clin Geriatr Med. 2020 Feb;36(1):1-12. doi: 10.1016/j.cger.2019.08.002. Epub 2019 Aug 24. PMID 31733690

DOCUMENTS (1):
  • Study Protocol (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT07068217/Prot_000.pdf